CLINICAL TRIAL: NCT04119817
Title: Clinical Study on the Effects of the Product Mucosave® on Gastrointestinal Discomfort and the Quality of Life in Healthy Volunteers
Brief Title: Effects of Mucosave® on Gastrointestinal Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUCOGASDISCOMFORT
Record Dates: First submitted 2019-09-19; First posted 2019-10-08 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Gastrointestinal Discomfort
Keywords: Gastrointestinal symptoms; Nausea; Heartburn; Reflux
MeSH Terms: conditions — Nausea; Heartburn; Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, double blind study
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mucosave® capsules (Experimental): 60 healthy volunteers taking 400 mg/day of Mucosave® capsules for a period of 8 weeks, once a day after dinner before going to bed.
  Interventions: Dietary Supplement: Mucosave® capsules
- Placebo (Placebo Comparator): 40 healthy volunteers taking capsules of placebo for a period of 8 weeks, once a day after dinner before going to bed.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mucosave® capsules — 400 mg/day of Mucosave® capsules for a period of 8 weeks, once a day.
  Arms: Mucosave® capsules
Dietary Supplement: Placebo — 400 mg/day of placebo capsules for a period of 8 weeks, once a day.
  Arms: Placebo

SUMMARY:
Gastrointestinal (GI) discomfort, which often includes gastroesophageal reflux disease (GERD) is a common disorder in healthy adults affecting 20% of people particularly women. The disorders related to GI discomfort usually have a huge impact on the quality of life. Current treatment for GERD are associated with side effects. In this study, researchers designed a randomized double-blind placebo-controlled trial to assess the effect of Mucosave® on the symptoms and quality of life of healthy adults with gastrointestinal discomfort. One hundred healthy subjects with GI discomfort were enrolled in the study and divided in two groups: 60 and 40 taking for 8 weeks Mucosave® (400 mg/day) or placebo (400 mg/day). To evaluate the effects of treatment, the questionnaires Gastrointestinal Quality of Life index (GIQLI) and GERD Symptom Assessment Scale (GSAS) were self-administered by participants before the beginning of period of supplementation (T0), after four weeks (T4) during the period of supplementation and after 8 weeks (T8) at the end of supplementation.

DETAILED DESCRIPTION:
Gastrointestinal (GI) discomfort is a common disorder in healthy adults with a prevalence of 20%, particularly affecting women. Gut health is gaining more interest nowadays for a variety of reasons including the well-established link between the body and mind via the brain-gut axis. As a result of this connection, GI discomfort is usually accompanied by psychosocial factors such as stress and mood disorders. The quality of life can therefore be reduced as there is also the occurrence of wide range of disorders, including abdominal pain, sense of fullness, nausea, sense of swelling, flatulence, bowel movements, constipation, eructation, heartburn and reflux. Gastroesophageal reflux disease (GERD), which is one of the most frequent causes of GI discomfort, is a chronic and relapsing disorder that occurs when the stomach content reflux into the esophagus. The condition is common in Western countries with a prevalence estimated to be about 10-20% while in Asia the occurrence is lower (5%) but is expected to increase in a near future. In the United State, 44% of the population report having GERD symptoms at least once a month and 20% at least once a week. Due to the accelerated pace of life in recent years with an important change in lifestyle, there is an increase in GERD incidence. Although GERD is not life threatening, it is characterized by important impairment in health related quality of life (HRQL) including a decrease in productivity comparable to that of other chronic diseases. In fact, HRQL has been demonstrated to be poorer in subjects with frequent upper gastrointestinal tract symptoms compared to those with no symptoms as measured by the Psychological General Well-Being Index . Beside the typical GERD symptoms like regurgitation and heartburn, impairment of quality of life include disturbed sleep, body pain, anxiety and unsatisfactory sex life. The reflux episodes can occur on daytime but nocturnal symptoms have an important influence on life quality and are associated to the complications of GERD. In addition, GERD symptoms impose a substantial cost on healthcare systems. Non pharmacological treatment of GERD include avoiding alcohol, coffee, smoking and reducing body weight. On the other hand, current pharmacological treatment primarily focuses on the use of proton pump inhibitors (PPIs) for the inhibition of gastric secretion. However, there is a persistence of troublesome GERD symptoms in 20-30% of patients after a daily treatment with a standard PPI dose. According to World Health Organization, about 80% of people in developing countries rely on herbal medicine as the first line of treatment. Natural plants present an interesting option for the management of gastrointestinal disorders. Opuntia ficus-indica (L.) also known as prickle pear is a tropical and subtropical plant usually growing in arid climates especially in the Mediterranean and Central America regions thanks to it special adaptative mechanism. In Sicily traditional medicine the plant's cladodes are used in the treatment of gastric ulcer. This traditional use has been confirmed by scientific studies, suggesting the mucoadhesion effect due to the polysaccharides content of cladodes. Wound healing properties are also attributed to Opuntia ficus-indica when topically applied on rats. On the other hand, Olea europea (Olive) is a mediterranean plant which leaves extract has been shown to prevent experimental formation of gastric lesions induced by stress. Other biological activities of olive leaves include anti-inflammatory and antioxidant thanks to its abundance in polyphenols. Furthermore, a significant correlation has recently been demonstrated between gastrointestinal discomfort and microbial dysbiosis. On this basis, the role of intestinal microbiota is emerging along with its importance as a new target for treatment.

A previous clinical study reported the efficacy and the safety for GERD treatment as a medical device based on sodium alginate/bicarbonate in combination with Mucosave®, a blend of extracts from Opuntia ficus-indica cladodes and Olea europea leaves . In this study, researchers performed a double-blinded randomized-controlled trial to assess the efficacy of Mucosave® as a sole primary therapy in healthy adults with gastrointestinal discomfort. The questionnaires used were the Gastrointestinal Quality of life Index (GIQLI) to evaluate the impact of the disorders on the quality of life and the GERD Symptom Assessment Scale (GSAS) designed to assess various aspects of GERD. Efficacy in reducing gastrointestinal disorders was also measured by the completion of a subjective daily diary.

Potential participants were subjected to a short medical visit and the inclusion and exclusion criteria were assessed and the possibility of inclusion in the study established. The study was performed in accordance with the principles of the Declaration of Helsinki. Written informed consent was obtained before subjects enrollment.

Calculation of the sample size The sample size was estimated considering as primary endpoint, the increase of the GIQLI score in the study period. Data in the literature show that healthy subjects have a GIQLI score variability value of 13.00 and in the present study included subjects with a GIQLI score not lower than 90.00. Therefore, considering a value (δ) of clinically relevant increase of the score equal to 10, an α value equal to 0.05 and a study power of 80%, 55 patients were required to carry out the experimentation. In order to guarantee the power, a possible abandonment rate of 8% was also considered, consequently a total number of 60 subjects supplied with Mucosave® is necessary to be guaranteed the endpoint of the study.

Screening and Randomisation Before enrollment subjects were asked to respond to the GIQLI and GSAS questionnaires with the aim to establish basal level score of participants.

Intervention Allocation of participants into the group supplied with Mucosave® or placebo was performed through computerized randomization. A total of 100 participants were enrolled. They were divided in two groups: 60 healthy volunteers taking 400 mg/day of Mucosave® capsules and 40 healthy volunteers taking capsules of placebo for a period of 8 weeks, once a day after dinner before going to bed. Mucosave® (Bionap srl, Italy) is a blend of two enriched extracts from Opuntia ficus-indica cladodes (32-35% w/w) and Olea europea (olive) leaves (23-25% w/w) with a total polyphenol amount of 3.7-4.3% as luteolin 7-O-glucoside with maltodextrin as support.

Assessment Compliance with test beverage consumption was self- recorded daily by participants in a diary. Subjects were reminded of the behavioural modalities related to the study: dosage of treatment and abstinence from taking anti-reflux drugs such as PPIs, histamine-2 blockers, agents facilitating motility or other antacids.

The primary endpoint of the study was defined as relief of gastrointestinal disorders evaluated by GIQLI and GSAS at the beginning (T0), after four weeks (T4) and eight weeks (T8) of supplementation period between the group of subjects supplied with Mucosave® and group supplied with placebo.

The Gastrointestinal Quality of Life Index (GIQLI) questionnaire contains 36 questions, each with 5 answers in the "Likert scale" style (technique for measuring the attitude): the range goes from 0 (always answer with letter "a") to 144 (always answer with letter "e"), according to the meaning "higher score, better quality of life". Patients with more severe gastro-intestinal disorders generally reach an average score corresponding to 45 points, compared to the median score 126 of healthy controls. Investigators analyzed answers and evaluated the scores only for the following disorders: abdominal pain, sense of fullness, sense of swelling, flatulence, eructation, bowel sounds, bowel movements, reflux, constipation, nausea and heartburn. Increase in scores corresponds to reduction of disorders.

GSAS is the most complete evaluation scale of gastrointestinal symptoms. The GSAS is a 15-item tool designed to evaluate various aspects including stress about gastrointestinal symptoms before and after treatments. It is a simple and easy to understand tool that can be administered in a relatively short time. GSAS is valid, stable and sensitive to changes in symptom over time.

At the same time each participant received a daily diary in which they found a few simple multiple choice questions, which helped the investigators to establish the individual degree of satisfaction of treatment. Each participant was asked to answer for the first 15 days of treatment with Mucosave® or placebo to the following questions: How are you today?, How are you compared to yesterday?, Have you had heartburn today?, have you had abdominal swelling today?, Have you had belching today?, Which symptoms were improved today?.

The symptom diaries and questionnaires were coded and anonymized. Codes were broken only after the raw data had been entered into the database.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women aged between 30 and 50 years;
* subjects able to read, to understand and to sign approval of informed consent;
* subjects not using food supplements for gastro-intestinal well-being;
* subjects available to continue own habitual diet;
* subjects without diagnosis of clinical diseases with relevant effects on the gastrointestinal system or visceral motility;
* subjects with reduced bowel movements defined as an average of > 1 and ≤ 3.5 stools per week in the last 6 months;
* subjects with BMI = 18-30 kg/m2;
* non-smoker subjects.

Exclusion Criteria:

* history of gastroesophageal surgery or endoscopic therapy due to severe erosive esophagitis;
* presence of Barrett's esophagus;
* subjects with uncontrolled or severe medical problems such as asthma, angina, hepatic or kidney diseases;
* subjects aged < 30 or > 50 years;
* presence of acute or chronic inflammatory processes requiring therapy;
* presence of acute or chronic coexisting diseases (cardiovascular, gastrointestinal, endocrinological, immunological, metabolic or any other condition that contraindicates, in the opinion of the investigators, the participation to the study);
* subjects taking drugs that, in the opinion of the investigator, may interfere with the objectives of the study or represent a safety risk or can confuse the interpretation of the study results including heartburn medication, probiotics and prebiotics;
* subjects that, in the opinion of the investigator, can be considered as potential participants, but for whatever reason are not able to respect the protocol of the study;
* pregnant or nursing women;
* subjects who cannot receive treatment with experimental drugs; subject participating in a recent experimental study (this must have been performed no less than 30 days prior to this study);
* subjects affected by neoplasms.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-09 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Evaluation of relief of gastrointestinal disorders with the Gastrointestinal Quality of Life Index (GIQLI) questionnaire. | 8 weeks
  The Gastrointestinal Quality of Life Index (GIQLI) questionnaire contains questions on gastrointestinal symptoms, each with 5 answers in the "Likert scale" style (technique for measuring the attitude), according to the meaning "higher score, better quality of life". The GIQLI is an appropriate, validated and potentially useful tool to assess health-related quality of life in clinical studies of patients with gastrointestinal disease.
  Each of the 36 items is scored on a five-point scale (0 to 4) denoting the burden of the particular symptom or dysfunction. The total score ranged from 0 (worst) to 144 (best quality of life) with higher scores representing better quality of life. Subscales can be summarized or averaged.
Evaluation of relief of gastrointestinal symptoms with the Gastroesophageal Reflux Disease Symptom Assessment Scale (GSAS): an evaluation scale of gastrointestinal symptoms. | 8 weeks
  GSAS is a 15-item tool designed to evaluate various aspects including stress about gastrointestinal symptoms before and after treatments. GSAS is a self-administered questionnaire that asks patients to report about the previous week for 15 specific symptoms: heartburn, a feeling of pressure inside chest, food coming back into mouth, an acid in mouth, frequent gurgling, feeling of lump in throat, nausea, burning pain in throat, bloating, belching, flatulence, feeling full after eating, bad breath, coughing, and hoarseness.
  Scoring of the GSAS distress subscale is based on the presence of the symptoms and their bother ratings. Specifically, patients first indicate whether they had the symptom in the past week. If they did not have the symptom, their score for the symptom is 0. If they did have the symptom, they then report how bothered they were by it on a 4-point scale (0 ? not at all, 1 ? somewhat, 2 ? quite a bit, 3 ? very much). Subscales can be summarized or averaged.

SECONDARY OUTCOMES:
Satisfaction of supplementation. | 15 days
  Each participant received a daily diary in which they found a few simple multiple choice questions, which helped the investigators to establish the individual degree of satisfaction of treatment. Each participant was asked to answer for the first 15 days of treatment with Mucosave® or placebo to the following questions: How are you today?, How are you compared to yesterday?, Have you had heartburn today?, have you had abdominal swelling today?, Have you had belching today?, Which symptoms were improved today?.
Intestinal microbiota investigation on stool samples | 8 weeks
  Each participant will collect a stool sample before and another at the end of period of supplementation for intestinal microbiota investigation .

CONTACTS AND LOCATIONS:
Overall Officials: Gioacchino Calapai, MD, Principal Investigator — Azienda Ospedaliera Universitaria "G Martino", Messina, Italy.
Locations (1):
- Gioacchino Calapai, Messina, Me, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buchwald-Werner S, Fujii H, Reule C, Schoen C. Perilla extract improves gastrointestinal discomfort in a randomized placebo controlled double blind human pilot study. BMC Complement Altern Med. 2014 May 27;14:173. doi: 10.1186/1472-6882-14-173. PMID 24885816
- [Background] Salehi M, Karegar-Borzi H, Karimi M, Rahimi R. Medicinal Plants for Management of Gastroesophageal Reflux Disease: A Review of Animal and Human Studies. J Altern Complement Med. 2017 Feb;23(2):82-95. doi: 10.1089/acm.2016.0233. Epub 2016 Dec 20. PMID 27996295
- [Background] Panahi Y, Khedmat H, Valizadegan G, Mohtashami R, Sahebkar A. Efficacy and safety of Aloe vera syrup for the treatment of gastroesophageal reflux disease: a pilot randomized positive-controlled trial. J Tradit Chin Med. 2015 Dec;35(6):632-6. doi: 10.1016/s0254-6272(15)30151-5. PMID 26742306
- [Background] Enck P, Dubois D, Marquis P. Quality of life in patients with upper gastrointestinal symptoms: results from the Domestic/International Gastroenterology Surveillance Study (DIGEST). Scand J Gastroenterol Suppl. 1999;231:48-54. doi: 10.1080/003655299750025264. PMID 10565623
- [Background] Alecci U, Bonina F, Bonina A, Rizza L, Inferrera S, Mannucci C, Calapai G. Efficacy and Safety of a Natural Remedy for the Treatment of Gastroesophageal Reflux: A Double-Blinded Randomized-Controlled Study. Evid Based Complement Alternat Med. 2016;2016:2581461. doi: 10.1155/2016/2581461. Epub 2016 Oct 12. PMID 27818697
- [Background] El-Serag H, Becher A, Jones R. Systematic review: persistent reflux symptoms on proton pump inhibitor therapy in primary care and community studies. Aliment Pharmacol Ther. 2010 Sep;32(6):720-37. doi: 10.1111/j.1365-2036.2010.04406.x. PMID 20662774
- [Background] Di Lorenzo F, Silipo A, Molinaro A, Parrilli M, Schiraldi C, D'Agostino A, Izzo E, Rizza L, Bonina A, Bonina F, Lanzetta R. The polysaccharide and low molecular weight components of Opuntia ficus indica cladodes: Structure and skin repairing properties. Carbohydr Polym. 2017 Feb 10;157:128-136. doi: 10.1016/j.carbpol.2016.09.073. Epub 2016 Sep 24. PMID 27987833
- [Background] Galati EM, Mondello MR, D'Aquino A, Miceli N, Sanogo R, Tzakou O, Monforte MT. Effects of Teucrium divaricatum Heldr. ssp. divaricatum decoction on experimental ulcer in rats. J Ethnopharmacol. 2000 Sep;72(1-2):337-42. doi: 10.1016/s0378-8741(00)00280-4. PMID 10967492
- [Background] Trombetta D, Saija A, Bisignano G, Arena S, Caruso S, Mazzanti G, Uccella N, Castelli F. Study on the mechanisms of the antibacterial action of some plant alpha,beta-unsaturated aldehydes. Lett Appl Microbiol. 2002;35(4):285-90. doi: 10.1046/j.1472-765x.2002.01190.x. PMID 12358689
- [Background] Dekanski D, Janicijevic-Hudomal S, Ristic S, Radonjic NV, Petronijevic ND, Piperski V, Mitrovic DM. Attenuation of cold restraint stress-induced gastric lesions by an olive leaf extract. Gen Physiol Biophys. 2009;28 Spec No:135-42. PMID 19893091
- [Background] El SN, Karakaya S. Olive tree (Olea europaea) leaves: potential beneficial effects on human health. Nutr Rev. 2009 Nov;67(11):632-8. doi: 10.1111/j.1753-4887.2009.00248.x. PMID 19906250
- [Background] Eypasch E, Wood-Dauphinee S, Williams JI, Ure B, Neugebauer E, Troidl H. [The Gastrointestinal Quality of Life Index. A clinical index for measuring patient status in gastroenterologic surgery]. Chirurg. 1993 Apr;64(4):264-74. German. PMID 8482141
- [Background] Revicki DA, Wood M, Wiklund I, Crawley J. Reliability and validity of the Gastrointestinal Symptom Rating Scale in patients with gastroesophageal reflux disease. Qual Life Res. 1998 Jan;7(1):75-83. doi: 10.1023/a:1008841022998. PMID 9481153
- [Background] Borgaonkar MR, Irvine EJ. Quality of life measurement in gastrointestinal and liver disorders. Gut. 2000 Sep;47(3):444-54. doi: 10.1136/gut.47.3.444. PMID 10940286
- [Background] Damiano A, Handley K, Adler E, Siddique R, Bhattacharyja A. Measuring symptom distress and health-related quality of life in clinical trials of gastroesophageal reflux disease treatment: further validation of the Gastroesophageal Reflux Disease Symptom Assessment Scale (GSAS). Dig Dis Sci. 2002 Jul;47(7):1530-7. doi: 10.1023/a:1015815102175. PMID 12141813
- [Background] Fass R. Symptom assessment tools for gastroesophageal reflux disease (GERD) treatment. J Clin Gastroenterol. 2007 May-Jun;41(5):437-44. doi: 10.1097/MCG.0b013e31802e849f. PMID 17450022
- [Background] Dupont HL. Review article: evidence for the role of gut microbiota in irritable bowel syndrome and its potential influence on therapeutic targets. Aliment Pharmacol Ther. 2014 May;39(10):1033-42. doi: 10.1111/apt.12728. Epub 2014 Mar 25. PMID 24665829